CLINICAL TRIAL: NCT02607059
Title: Epidemiologic Registry of Patients Diagnosed With Acute Myeloid Leukemia (PETHEMA LMA 2015)
Brief Title: Epidemiologic Registry PETHEMA LMA 2015
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: LAM 2015
Record Dates: First submitted 2015-10-13; First posted 2015-11-17 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: AML
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Registry

SUMMARY:
Epidemiologic and retrospective multicenter registry of all patients diagnosed with de novo or secondary acute myeloid leukemia (AML) in the PETHEMA Group institutions. This study is a non-interventional research regarding diagnosis and therapeutic approach

DETAILED DESCRIPTION:
To perform this registry, every patient diagnosed with AML in the participant institutions, regardless type of AML and treatment administered, must be reported. It will be required to registry the main characteristics of the patients and AML at diagnosis, as cytomorphologic, immunophenotypic, and cytogenetic results, according to the habitual practice of the centers. The treatment which has been administered by every center of the PETHEMA Group, even when it is considered as supportive care, and evolution of the disease will also be reported (relapse o death). PETHEMA Group will input all the reported information in data bases

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with acute myeloid leukemia

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
characteristics of the patients diagnosed of AML | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital La Fe, Valencia, Spain

REFERENCES:
- [Derived] Labrador J, Martinez-Cuadron D, Boluda B, Serrano J, Gil C, Perez-Simon JA, Bernal T, Bergua JM, Martinez-Lopez J, Rodriguez-Medina C, Vidriales MB, Garcia-Boyero R, Algarra L, Polo M, Sayas MJ, Tormo M, Alonso-Dominguez JM, Herrera P, Lavilla E, Ramos F, Amigo ML, Vives-Polo S, Rodriguez-Macias G, Mena-Duran A, Perez-Encinas MM, Arce-Fernandez O, Cuello R, Sanchez-Garcia J, Gomez-Casares MT, Chillon MC, Calasanz MJ, Ayala R, Rodriguez-Veiga R, Barragan E, Montesinos P; PETHEMA Group. Evolving patterns and clinical outcome of genetic studies performed at diagnosis in acute myeloid leukemia patients: Real life data from the PETHEMA Registry. Cancer. 2024 Oct 15;130(20):3436-3451. doi: 10.1002/cncr.35431. Epub 2024 Jun 19. PMID 38896056
- [Derived] Martinez-Cuadron D, Megias-Vericat JE, Serrano J, Martinez-Sanchez P, Rodriguez-Arboli E, Gil C, Aguiar E, Bergua J, Lopez-Lorenzo JL, Bernal T, Espadana A, Colorado M, Rodriguez-Medina C, Lopez-Pavia M, Tormo M, Algarra L, Amigo ML, Sayas MJ, Labrador J, Rodriguez-Gutierrez JI, Benavente C, Costilla-Barriga L, Garcia-Boyero R, Lavilla-Rubira E, Vives S, Herrera P, Garcia-Belmonte D, Herraez MM, Vasconcelos Esteves G, Gomez-Roncero MI, Cabello A, Bautista G, Balerdi A, Mariz J, Boluda B, Sanz MA, Montesinos P. Treatment patterns and outcomes of 2310 patients with secondary acute myeloid leukemia: a PETHEMA registry study. Blood Adv. 2022 Feb 22;6(4):1278-1295. doi: 10.1182/bloodadvances.2021005335. PMID 34794172